CLINICAL TRIAL: NCT03427450
Title: Harvest of Circulating Tumor Cells (CTCs) From Patients With Metastatic Breast Cancer (MBC) Using the Parsortix™ PC1 System
Brief Title: Harvest of CTCs From MBC Patients Using the Parsortix™ PC1 System
Acronym: HOMING
Status: Completed | Type: Observational
Sponsor: Angle plc (Industry)
Responsible Party: Sponsor
Other Study IDs: ANG-002
Record Dates: First submitted 2018-01-31; First posted 2018-02-09 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Healthy Volunteers; Breast Cancer, Metastatic
Keywords: circulating tumor cells; liquid biopsy; microfluidics
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cytology slides Her2 FISH slides mRNA cDNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Healthy Volunteers (Controls): A control population of healthy volunteers (HVs) consisting of women with no prior/current history of cancer and no known history of breast disease (the information obtained from the HVs may be 'self-reports', as complete medical records may not be available at the enrolling site for these control subjects), and with a broadly similar age range to the cancer patient study population. All eligible and consenting subjects will have blood draw.
  Interventions: Diagnostic Test: Blood draw
- MBC Patients (Cancers): Women with either newly diagnosed metastatic breast cancer who are about to start a new line of therapy of any type for the treatment and/or management of their disease or those with currently progressive or recurrent disease (as determined by any means) will be eligible for enrollment into the cancer population. All eligible and consenting subjects will have blood draw.
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — Blood collected will be processed on Parsortix PC1 system for capture and harvest of circulating tumor cells to be used in subsequent evaluations.

SUMMARY:
The purpose of this clinical study is to demonstrate that the Parsortix™ PC1 system enables the capture and harvest of circulating tumor cells (CTCs) from the peripheral blood of patients with metastatic breast cancer (MBC) and not from healthy volunteers (HVs). The study is also designed to demonstrate that the CTCs harvested by the Parsortix PC1 system from MBC patients can be used effectively for different types of evaluations (e.g. cytopathology, FISH, qPCR, RNAseq, etc.).

This is an investigational study. The Parsortix PC1 system is not FDA approved and is currently being used for research purposes only.

DETAILED DESCRIPTION:
Approximately 200 evaluable MBC patients (either newly diagnosed or patients with progressive/recurrent disease who are about to start a new line of therapy for the treatment of their disease) and 200 evaluable healthy volunteer (HV) subjects (healthy women with no history of cancer) will be enrolled at a minimum of three (3) US based clinical sites. Each subject will have information about their age race/ethnicity, height and weight, menopausal status, smoking status, pregnancy and/or nursing status, and a brief medical history captured at the time of enrollment. Blood will be drawn from each subject into three different EDTA tubes (minimum of ~7mL up to a maximum of ~23mL of whole blood) specifically for the purposes of this study. One of the blood tubes collected will be used for a complete blood count (CBC) with differential testing, while the other two tubes of blood will be processed on the Parsortix PC1 system for the capture and harvest of CTCs. The cells harvested from one of the blood tubes will be deposited onto a glass slide and automated Wright-Giemsa staining will be done to allow for identification of CTCs based on their cytologic features (e.g. size, shape, nuclear to cytoplasmic ratio, chromatin structure, etc.) by an expert cytopathologist. The cells harvested from the remaining blood tube will be used for one of three different evaluations: Fluorescence in-situ hybridization (FISH) for evaluation of Her-2/neu gene amplification, quantitative reverse-transcriptase real-time PCR (qRT-PCR) for evaluation of cancer related gene expression, or whole transcriptome sequencing (RNAseq) for determination of the expression patterns of breast cancer related genes.

ELIGIBILITY:
MBC Patient Inclusion Criteria

* Female >=22 years of age;
* Documented evidence of metastatic breast cancer (i.e. primary tumor histopathology of breast cancer and documented evidence of distant sites of metastasis by imaging, biopsy, or other means) that is either newly diagnosed or currently progressing / recurrent (disease progression / recurrence may be determined by any means, including RECIST v1.1 criteria, physical signs and symptoms, rising tumor markers, physician determination, etc.);

  * If newly diagnosed, have not yet started a new line of therapy of any type (e.g. hormonal, cytotoxic, targeted, etc.) for the treatment and/or management of their metastatic breast cancer;
  * If progressing or recurrent, any number of prior hormonal therapies, chemotherapies and/or biological/targeted therapies are allowed;
* Willing and able to provide informed consent and agree to complete all aspects of the study.

MBC Patient Exclusion Criteria

* Female subjects <=21 years old or male subjects;
* Concurrent other malignancies (except for a second primary breast cancer);
* Less than seven days since last administration of a cytotoxic agent;
* Unwilling or unable to provide informed consent or high risk that subject may not comply with protocol requirements.

HV Inclusion Criteria

* Females >=22 years of age;
* No known fever or active infections at the time of the blood collection;
* No known current diagnosis of acute inflammatory disease or chronic inflammation;
* No known current and/or prior history of malignancy, excluding skin cancers (squamous cell or basal cell);
* Willing and able to provide informed consent and agree to complete all aspects of the study.

HV Exclusion Criteria

* Female subjects <=21 years old or male subjects;
* Known illness at the time of the blood collection;
* Known current and/or prior history of malignancy, excluding skin cancers (squamous cell or basal cell);
* Unwilling or unable to provide informed consent or high risk that subject may not comply with protocol requirements (e.g. due to health and/or participation in other research studies).

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers: Female subjects at outpatient clinics whom a delegated physician and/or study coordinator believe may be eligible for the study will be approached by the delegated physician and/or study coordinator during their scheduled gynecology appointment or, if they are accompanying a breast cancer patient, during the scheduled appointment of the individual they are accompanying.
  Metastatic Breast Cancer Patients: Eligible female subjects at outpatient clinics and/or under the care of investigators at the participating medical centers will be prospectively identified by the site principal investigator, sub-investigators, nurses and/or study coordinator.
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of CTC | 1 day (At time of blood draw)
  Determine the proportion of MBC patients and healthy volunteers (HVs or controls) that have one or more observable CTCs (as determined by a qualified pathologist using cytological evaluation of Wright-Giemsa stained slides) harvested from their peripheral blood using the Parsortix PC1 system.

SECONDARY OUTCOMES:
CTC Enumeration | 1 day (At time of blood draw)
  Quantify the number of observable CTCs (as determined by a qualified pathologist using cytological evaluation of Wright-Giemsa stained slides) harvested from the peripheral blood of each MBC patient and healthy volunteer (HV or control) and summarize separately for each group.

OTHER OUTCOMES:
Her2 FISH Evaluation | 1 day (At time of blood draw)
  Demonstrate that CTCs harvested from peripheral blood of MBC patients by the Parsortix PC1 system and deposited onto slides can be evaluated by fluorescence in-situ hybridization (FISH) for Her-2/neu gene amplification.
qPCR Evaluation | 1 day (At time of blood draw)
  Demonstrate that CTCs harvested from peripheral blood of MBC patients by the Parsortix PC1 system and deposited into an RNA preservation/lysis buffer can be evaluated using qPCR for analysis of cancer related gene expression.
RNAseq Evaluation | 1 day (At time of blood draw)
  Demonstrate that CTCs harvested from peripheral blood of MBC patients by the Parsortix PC1 system and deposited into an RNA preservation/lysis buffer can be evaluated using whole genome sequencing (RNAseq) for determination of the expression patterns of breast cancer related genes.

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PhD, Principal Investigator — UT MD Anderson Cancer Center
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Rochester Medical Center Wilmot Cancer Institute, Rochester, New York
  - UT MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu L, Mao X, Imrali A, Syed F, Mutsvangwa K, Berney D, Cathcart P, Hines J, Shamash J, Lu YJ. Optimization and Evaluation of a Novel Size Based Circulating Tumor Cell Isolation System. PLoS One. 2015 Sep 23;10(9):e0138032. doi: 10.1371/journal.pone.0138032. eCollection 2015. PMID 26397728
- [Background] Hvichia GE, Parveen Z, Wagner C, Janning M, Quidde J, Stein A, Muller V, Loges S, Neves RP, Stoecklein NH, Wikman H, Riethdorf S, Pantel K, Gorges TM. A novel microfluidic platform for size and deformability based separation and the subsequent molecular characterization of viable circulating tumor cells. Int J Cancer. 2016 Jun 15;138(12):2894-904. doi: 10.1002/ijc.30007. Epub 2016 Feb 26. PMID 26789903
- [Result] Cohen EN, Jayachandran G, Moore RG, Cristofanilli M, Lang JE, Khoury JD, Press MF, Kim KK, Khazan N, Zhang Q, Zhang Y, Kaur P, Guzman R, Miller MC, Reuben JM, Ueno NT. A Multi-Center Clinical Study to Harvest and Characterize Circulating Tumor Cells from Patients with Metastatic Breast Cancer Using the Parsortix(R) PC1 System. Cancers (Basel). 2022 Oct 26;14(21):5238. doi: 10.3390/cancers14215238. PMID 36358657